#### **B.** Braun Medical Inc.

#### HC-G-H-1601

A Phase 4, Open-Label, Single-Dose, Parallel-Group Study to Evaluate the Safety of 1 g of Cefazolin in Pediatric Subjects With a Weight of at Least 25 kg but Less Than 60 kg Scheduled for Surgery and the Safety of 2 g of Cefazolin in Pediatric Subjects with a Weight of at Least 60 kg Scheduled for Surgery

#### 15NOV2017

Final Statistical Analysis Plan

Version 1.0

Prepared by:

PPD 3900 Paramount Parkway Morrisville, NC 27560 USA

# TABLE OF CONTENTS

| LIST | OF ABBREVIATIONS | . 4 |
|------|------------------------------------------------------|-----|
| 1. | INTRODUCTION | . 5 |
| 2. | OBJECTIVES | . 5 |
| 3. | INVESTIGATIONAL PLAN | . 6 |
| 3.1. | OVERALL STUDY DESIGN AND PLAN | . 6 |
| 3.2. | STUDY ENDPOINTS | |
| 3.3. | Treatments | . 7 |
| 3.4. | Dose Adjustment/Modifications | |
| 4. | GENERAL STATISTICAL CONSIDERATIONS | . 7 |
| 4.1. | SAMPLE SIZE | . 8 |
| 4.2. | RANDOMIZATION, STRATIFICATION, AND BLINDING | . 8 |
| 4.3. | Analysis Sets | . 9 |
| 4 | 3.1. Safety | . 9 |
| 4 | 3.2. Pharmacokinetic | . 9 |
| 5. | SUBJECT DISPOSITION | . 9 |
| 5.1. | DISPOSITION | . 9 |
| 5.2. | PROTOCOL DEVIATIONS | |
| 6. | DEMOGRAPHICS AND BASELINE CHARACTERISTICS | 10 |
| 6.1. | Demographics | 10 |
| 6.2. | MEDICAL HISTORY | 10 |
| 7. | TREATMENTS AND MEDICATIONS | 10 |
| 7.1. | PRIOR AND CONCOMITANT MEDICATIONS | 10 |
| 7.2. | MEDICAL OR SURGICAL TREATMENT PROCEDURES | |
| 7.3. | Surgery | 11 |
| 7.4. | STUDY TREATMENTS | 11 |
| 8. | SAFETY ANALYSIS | 11 |
| 8 1 | Adverse Events | 11 |
| 8. | 1.1. Incidence of Adverse Events | 12 |
| 8. | 1.2. Relationship of Adverse Events to Study Drug | |
| 8. | 1.3. Severity of Adverse Event | |
| 8. | 1.4. Serious Adverse Events | |
| 8. | 1.5. Adverse Events Leading to Early Discontinuation | 13 |
| 8.2. | CLINICAL LABORATORY EVALUATIONS | |
| 8.3. | VITAL SIGN MEASUREMENTS | 14 |
| 8.4. | PHYSICAL EXAMINATION | 15 |
| 8.5. | ELECTROCARDIOGRAPH | 15 |
| 8.6. | OTHER SAFETY DATA | 15 |
| 9. | PHARMACOKINETICS | 16 |

| 10. | INTERIM ANALYSIS | 16 |
|------|------------------------------------------------------|----|
| 11. | REFERENCES | 16 |
| 12. | APPENDICES | 17 |
| 12.1 | . SCHEDULE OF STUDY PROCEDURES | 17 |
| | . TABLE, LISTING, AND FIGURE SHELL TABLE OF CONTENTS | |

#### **List of Abbreviations**

AE adverse event
CRF case report form
CSR clinical study report
ECG electrocardiogram

FDA Food and Drug Administration

IV intravenous

LAR legally authorized representative

MedDRA Medical Dictionary for Regulatory Activities

PK pharmacokinetic(s) PT preferred term

SAE serious adverse event SOC system organ class

USP United States Pharmacopeia WHO World Health Organization

#### 1. Introduction

Cefazolin for Injection United States Pharmacopeia (USP) and Dextrose Injection USP is a sterile, nonpyrogenic, single-use, packaged combination of Cefazolin Sodium USP (lyophilized) and sterile iso-osmotic diluent (i.e., Dextrose Injection USP) in the DUPLEX® sterile container and are supplied as a lyophilized form equivalent to either 1 g or 2 g of cefazolin.

Currently, cefazolin is a standard of care for perioperative infection prophylaxis in pediatric patients and is administered in a wide variety of surgical procedures. Older children and adolescents may benefit from the availability of a fixed-dose system for the prophylactic administration of cefazolin.

This study is a post-marketing requirement established by the Food and Drug Administration (FDA) as part of the Pediatric Research Equity Act to evaluate the safety of cefazolin in children aged 10 to 17 years (inclusive) receiving weight-based 1 g or 2 g of cefazolin intravenously over 30 minutes delivered via the DUPLEX drug delivery system for surgical prophylaxis.

This document outlines the statistical methods to be implemented during the analysis of data collected within the scope of B. Braun Medical Inc., protocol HC-G-H-1601 version 2.0 (A Phase 4, Open-Label, Single-Dose, Parallel-Group Study to Evaluate the Safety of 1 g of Cefazolin in Pediatric Subjects With a Weight of at Least 25 kg but Less than 60 kg Scheduled for Surgery and the Safety of 2 g of Cefazolin in Pediatric Subjects With a Weight of at Least 60 kg Scheduled for Surgery), dated 24 March 2017. The purpose of this plan is to provide specific guidelines for which the analysis will proceed. Any deviations from these guidelines will be documented in the clinical study report (CSR). The analyses described in this plan are considered a priori, in that they have been defined prior to database lock. Any analyses performed subsequent to database lock will be considered post-hoc and exploratory. Post-hoc analyses will be identified in the CSR.

# 2. Objectives

The primary objective of this study is to evaluate the safety of a single 30-minute infusion of a weight-based dose of cefazolin (1 g or 2 g) in pediatric subjects between 10 and 17 years of age (inclusive) scheduled for surgery.

The secondary objective of this study is to determine the cefazolin plasma concentrations following a single 30-minute infusion of a weight-based dose of cefazolin (1 g or 2 g) in pediatric subjects between 10 and 17 years of age (inclusive) scheduled for surgery.

#### 3. Investigational Plan

#### 3.1. Overall Study Design and Plan

This is a Phase 4, open-label, single-dose, parallel-group, multicenter, safety study of cefazolin (1 g or 2 g) in pediatric subjects between 10 and 17 years of age (inclusive) scheduled for surgery. This study will be conducted at approximately 5 study sites (to a maximum of 15 sites) in the United States.

Approximately 110 subjects will be enrolled and assigned to 1 of the 2 dose groups in a 1:1 ratio (55 subjects in each group). Subjects with a weight of at least 25 kg but less than 60 kg will receive a single dose of 1-g cefazolin. Subjects with a weight of at least 60 kg will receive a single dose of 2-g cefazolin. Dose groups will not be balanced by age or gender. Additional subjects may be enrolled if necessary to ensure at least 50 evaluable subjects with complete safety data per dose group complete the study.

The study consists of a Screening Period of up to 30 days, a Treatment Period on Day 1 (day of surgery), and a Follow-up Period including a visit on Day 8 (±1 day). The maximal study duration for an individual subject will be 39 days. Safety will be assessed by monitoring adverse events (AEs), physical examination, vital signs, electrocardiographs (ECGs), and clinical laboratory tests. In addition, 4 pharmacokinetic (PK) samples will be obtained in a subset of approximately 40 subjects to determine the cefazolin plasma concentrations in this population. A minimum of ten of these 40 subjects are planned to be in the 10 to 13-year-old age bracket.

The schedule of study procedures is presented in Appendix 12.1.

#### 3.2. Study Endpoints

The primary endpoints are:

- Type and incidence of AEs
- Physical examination
- Vital signs (systolic and diastolic blood pressure, pulse, respiratory rate, and oral body temperature)
- ECGs
- Clinical laboratory tests (hematology and clinical chemistry)

The PK endpoint is:

• PK plasma concentrations of cefazolin

The PK analysis will be detailed in a separate document.

#### 3.3. Treatments

A peripheral venous catheter will be placed for all subjects before the start of the study drug administration for the intravenous (IV) infusion of the cefazolin and dextrose solution. Subjects with a weight of at least 25 kg but less than 60 kg will receive 1-g cefazolin. Subjects with a weight of at least 60 kg will receive 2-g cefazolin. After reconstitution, the solution will be administered over 30 minutes through an infusion line by using an infusion pump on Day 1 (day of surgery) for surgery prophylaxis. The study drug administration will begin 0.5 to 1 hour prior to the start of surgery and following institution guidelines.

### 3.4. Dose Adjustment/Modifications

If surgery is unexpectedly extended beyond the 3-hour limit, additional doses of study drug are permitted according to institutional guidelines. For subjects who consent to participate in PK sampling, best efforts will be made to obtain the 3-hour and possibly the 4-hour PK samples prior to administration of the additional dose of study drug. PK sample collection will not continue after administration of an additional dose of study drug. In this case, subjects from whom a 3-hour PK sample is obtained prior to administration of the additional dose are considered PK completers.

#### 4. General Statistical Considerations

Statistical analysis of the Safety and PK sets will be performed using SAS® software (SAS Institute Inc., Cary, North Carolina) version 9.3 or later. Descriptive statistics will be presented for all safety parameters. Continuous variables will be summarized by treatment group using the mean, SD, median, minimum value, and maximum value. Categorical variables will be summarized using frequency counts and percentages.

No inferential statistical analysis will be performed.

Baseline will be defined as the values obtained at Screening.

All data collected during the study will be analyzed and reported unless stated otherwise. No algorithm for missing data imputation will be employed.

If there are repeated measurements at a time point, the original scheduled measurement at that time point will be used in the summary tables. If the original scheduled measurement at that time point is missing, the next available repeated measurement will be used in the summary tables.

Unscheduled results will not be included in the summary tables except for determining Baseline, but will be presented in data listings.

# 4.1. Sample Size

Approximately 110 subjects (males and females) will be enrolled in this study. This sample size was determined based on the requirement of the FDA as part of the Pediatric Research Equity Act to evaluate the safety of a single dose of cefazolin for surgical prophylaxis in 100 pediatric subjects using the dose equivalent to 2-g cefazolin exposure in adults.

Additional subjects may be enrolled if necessary to ensure at least 50 evaluable subjects with complete safety data per dose group complete the study.

Approximately 40 subjects (males and females across both dose groups) will be enrolled in the PK subgroup. This sample size was determined using model-based simulations designed to explore both the number of subjects needed and the optimal times at which to obtain PK samples from those subjects. The previously-developed population PK model (Trang et al 2014) was employed using permutations introduced empirically to approximate potential PK differences in children enrolled in this study. Specifically, the previous population PK analysis found that pediatric surgical patients had, on average, 32% slower cefazolin clearance than healthy adult volunteers. The model-based simulations assessed how many subjects would be required to adequately capture the "true" difference in clearance between pediatric surgical subjects and healthy adults if the underlying difference was either greater than previous observation (i.e., a 50% decrease in clearance) or less than the previous observation (25%, 10%, or 0% difference). A range of sample sizes and PK sampling schemes were evaluated. Note that optimal sampling schemes were first identified using a multiple linear regression approach and then verified using the model-based simulations.

The results of the model-based simulation analyses indicated that a sample size of 40 subjects, each of which provides 4 blood samples for cefazolin assay at times of 0.5 to 1.0 hours, 2.0 hours, 3.0 hours, and 4.0 hours after the start of the cefazolin infusion, would be expected to provide adequate power to detect the true difference in clearance between pediatric surgical subjects and healthy adult volunteers.

A minimum of 10 of the 40 PK subjects are planned to be in the 10- to 13-year-old age bracket to ensure adequate representation of that age bracket in the refined population PK model.

Additional subjects maybe enrolled if necessary to ensure complete PK data from at least 40 subjects.

### 4.2. Randomization, Stratification, and Blinding

This is an open-label, non-randomized study.

#### 4.3. Analysis Sets

#### **4.3.1.** Safety

The safety analysis set will consist of all subjects who received any study drug. All analyses using the safety analysis set will group subjects according to treatment actually received. This analysis set will be used for the primary analysis.

#### 4.3.2. Pharmacokinetic

The PK analysis set will consist of all subjects from whom at least one measurable concentration PK sample is obtained.

### 5. Subject Disposition

## 5.1. Disposition

Subject disposition will be summarized for the safety analysis set and presented by treatment. The summary table includes the number and percentage of subjects who completed the study, subjects who discontinued from the study, subjects in the safety analysis set, and subjects in the PK set. All percentages will be based on the number of subjects in the safety analysis set.

The reasons for study discontinuation will also be summarized in this table. The reason for study discontinuation may include any of the following: protocol violation, noncompliance with the protocol, serious AE (SAE), intolerable AE, lost to follow-up, pregnancy, subject withdrew consent, legally authorized representative (LAR) withdrew consent, or investigator decision.

Subject disposition data will be presented in a listing. Subject informed consent and assent data will be presented in a listing.

Admission criteria deviations will be presented in a listing.

Subjects excluded from any analysis population will be presented in a listing.

#### 5.2. Protocol Deviations

Protocol deviations are defined in the Study Deviation Rules document. All protocol deviations will be recorded in a clinical trial management system and reviewed. Any deviations deemed CSR reportable after review will be presented in a data listing.

#### 6. Demographics and Baseline Characteristics

## 6.1. Demographics

A summary of demographics and baseline information will be presented by treatment and overall. This summary will be presented for both the safety analysis set and the PK analysis set. The demographic characteristics consist of age (years), sex, race, and ethnicity. The baseline characteristics consist of baseline height (cm) and baseline weight (kg).

A subject's age in years will be calculated using the date of the informed consent and date of birth. Age (years), baseline height (cm), and baseline weight (kg). The number and percentage of subjects by age category (>=10 to <=13, >13 to <=17), sex (Male, Female), race (White, Black or African American, Asian, American Indian or Alaska Native, Native Hawaiian or Other Pacific Islander, and Other) and ethnicity (Hispanic or Latino, Not Hispanic or Latino), will also be reported. Percentages will be based on the total number of subjects in the analysis set.

Subject demographic and baseline characteristics will be presented in a listing.

## 6.2. Medical History

A complete medical history will be taken at the Screening visit. Medical history will be updated prior to surgery on Day 1 of the study. Medical history data will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) dictionary and presented in a listing.

#### 7. Treatments and Medications

#### 7.1. Prior and Concomitant Medications

The use of any medication (e.g., prescription, herbal, over-the-counter medication[s] or dietary supplements) known to interact with cefazolin within 5 days prior to the study drug administration until completion of the follow-up visit is prohibited. Concomitant use of probenecid is also prohibited for this period. Any concomitant medications taken during conduct of the study (from Screening through completion of follow-up) will be recorded in the case report form (CRF), as well as any changes in concomitant medications. This will include all prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications. All medications will be coded according to the World Health Organization drug dictionary (WHODrug version 01DEC2016).

Prior and concomitant medications will be presented in a listing.

#### 7.2. Medical or Surgical Treatment Procedures

The occurrence of any medical or surgical treatment procedure (aside from the primary surgery associated with cefazolin treatment) during the conduct of the study (from Screening through completion of follow-up) will be recorded in the CRF. All procedures will be coded according to the MedDRA dictionary, version 19.1. Medical and surgical procedures will be presented in a listing.

#### 7.3. Surgery

Details of the surgery associated with cefazolin treatment will be collected in the CRF. Surgery data will be presented in a listing.

#### 7.4. Study Treatments

Dosing details, including location of infusion catheter, whether any interruption of the infusion occurred with relevant dates and times, and volume of dose administered will be recorded in the CRF for the planned dose as well as any supplemental doses. This data will be presented in a listing.

# 8. Safety Analysis

#### 8.1. Adverse Events

An AE is defined as any untoward medical occurrence in a subject enrolled into this study regardless of its causal relationship to study drug. In addition to subject observations, AEs identified from any study data (e.g., laboratory values, physical examination findings, vital sign changes) or identified from review of other documents that are relevant to subject safety will be documented on the AE page in the CRF.

An AE is treatment emergent if it is not present before exposure to study drug or the event worsens in either intensity or frequency after exposure to study drug. Only treatment-emergent AEs that were not present at Screening or described in medical history will be reported in the CRF and included in summary tables and listings.

In all summary tables, system organ class (SOC) is displayed in descending order of frequency for "Total", then alphabetically. Preferred term (PT) is displayed in descending order of frequency for "Total", then alphabetically within SOC. Percentages will be based upon the number of subjects in the safety analysis set overall and within each treatment. At each level of subject summarization, a subject with 2 or more AEs will be counted only once in that level using the most severe event (for the severity table) or the most related event (for the relationship to study drug table).

The MedDRA version 19.1 will be used to code all AEs.

All analyses of AEs will be conducted using the safety analysis set.

#### 8.1.1. Incidence of Adverse Events

Summaries of the number and percentage of subjects with at least one AE will be provided by treatment group and overall. AEs will be presented by SOC and PT. At each level of subject summarization, a subject is counted once if the subject reported one or more events.

All AEs will be presented in a listing.

#### 8.1.2. Relationship of Adverse Events to Study Drug

A summary of AEs by relationship to study drug will be presented in a table by incidence of occurrence. The investigator will provide an assessment of the relationship of the event to the study drug. The possible relationships are "Unrelated", "Possible", "Probable", and "Definite". In the AE relationship table, if a subject reports multiple occurrences of the same AE, only the most closely related occurrence will be presented. If a subject has the relationship missing for all occurrences of the same AE, then the relationship will be presented in the summary tables as "Missing". AEs that are missing a relationship will be presented in the data listing with a missing relationship.

#### 8.1.3. Severity of Adverse Event

A summary of AEs by severity will be presented in a table. The severity that will be presented represents the most extreme severity captured on the CRF page. The possible severities are "Mild," "Moderate," and "Severe." In the AE severity table, if a subject reported multiple occurrences of the same AE, the subject will be counted only once for the most severe occurrence. AEs that are missing severity will be presented in tables as "Missing" and will be presented in the data listing with a missing severity.

#### 8.1.4. Serious Adverse Events

The seriousness of an AE should be assessed by the Investigator independently from the severity of the AE. An SAE is an event that results in death, is immediately life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect. Important medical events that may not result in death, be life threatening, or require hospitalization may be considered SAEs when, based upon appropriate medical judgment, they may jeopardize the

subject or may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

The SAEs will be listed.

#### 8.1.5. Adverse Events Leading to Early Discontinuation

All AEs leading to study discontinuation will be listed. An AE will be considered to have led to study discontinuation if the AE's identifier is listed on a subject's study completion form and that subject has given "Serious AE" or "Intolerable AE" as the primary reason for discontinuation.

#### 8.2. Clinical Laboratory Evaluations

Laboratory tests except for screening procedures will be performed by the central laboratory. Screening laboratory tests should be performed within 30 days of Day 1 and can be the same tests as assessed for surgical clearance. Screening laboratory tests will be performed at local laboratories. Aliquots of the serum and plasma collected at Screening will be sent to the central laboratory for replicate analysis and will serve as the baseline laboratory values. Blood samples for clinical laboratory assessments (hematology and chemistry) will be collected at Screening, Presurgery, Postsurgyre, and Follow-up. Urine samples for pregnancy testing will be collected at Screening and Presurgery.

All summaries will be based on SI units. In the event that the aliquots provide to the central lab cannot be used to determine the baseline lab values, local lab values will be entered into the CRF. These values will be converted to the same units as the central lab values.

The following laboratory analyses will be performed:

| Hematology | Clinical Chemistry |
|---|---|
| Hemoglobin | Alanine aminotransferase |
| <ul> <li>Hematocrit</li> </ul> | <ul> <li>Albumin</li> </ul> |
| <ul> <li>Mean corpuscular volume</li> </ul> | <ul> <li>Alkaline phosphatase</li> </ul> |
| <ul> <li>Mean corpuscular hemoglobin</li> </ul> | <ul> <li>Aspartate aminotransferase</li> </ul> |
| <ul> <li>Mean corpuscular hemoglobin</li> </ul> | <ul> <li>Blood urea nitrogen</li> </ul> |
| concentration | <ul> <li>Serum creatinine</li> </ul> |
| • Platelets | <ul> <li>Total bilirubin</li> </ul> |
| <ul> <li>Red blood cell</li> </ul> | • Sodium |
| <ul> <li>White blood cell with</li> </ul> | <ul> <li>Potassium</li> </ul> |
| differential count | <ul> <li>Chloride</li> </ul> |
| | <ul> <li>Bicarbonate</li> </ul> |
| | • Glucose |
| | • Uric acid |
| | • Calcium |
| | <ul> <li>Phosphate</li> </ul> |
| | <ul> <li>Total protein</li> </ul> |
| | <ul> <li>Creatine phosphokinase</li> </ul> |
| | Lactic acid dehydrogenase |

Baseline is defined in section 4.

Summary tables presenting observed values and changes from baseline will be presented for hematology and clinical chemistry results with numeric values by treatment and overall for subjects in the safety analysis set.

All clinical laboratory test results (including urine pregnancy) will be presented in the data listings sorted by subject, laboratory test, and sample collection date/time. For hematology and clinical chemistry, values that are outside of the normal reference range will be flagged in the listings.

#### 8.3. Vital Sign Measurements

Vital signs (including blood pressure [systolic and diastolic], pulse, body temperature, and respiratory rate) will be measured and assessed at Screening, Day 1, and at the follow up visit on Day 8 (±1 day). Pre-surgery vital sign measurements should be obtained within approximately 30 minutes before the start of study drug administration. Time points for vital sign measurements on Day 1 are pre-surgery, 15 minutes [±5 minutes], 0.5 to 1.0 hour, and 3.0 hours [±15minutes] after the start of the study drug infusion, and after surgery.

A summary table presenting observed values and changes from baseline will be presented for vital sign data, including systolic blood pressure (mmHg), diastolic blood pressure (mmHg), temperature (°C), pulse (beats/minute), and respiration (breaths/minute), by treatment and overall for subjects in the safety analysis set.

All vital sign data (both observed and change from baseline) will be presented in a listing.

#### 8.4. Physical Examination

A complete physical examination will be performed at Screening. The complete physical examination includes an assessment of general appearance and a review of systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, and respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, neurologic, and psychiatric systems).

A brief physical examination will be performed both before and after dosing on Day 1 and at the follow up visit.

Abnormal physical examination findings will be listed.

# 8.5. Electrocardiograph

Electrocardiographs will be performed at Screening and post-surgery. Clinical review and assessment of cardiac rhythm, conduction, waveform morphology and ECG interval duration will be performed at the study site, as close as possible to the time an ECG was obtained, by the investigator or his/her designee.

A summary table presenting observed values and changes from baseline will be presented for ECG data, including heart rate (bpm), PR Interval (msec), QRS Duration (msec), QT Interval (msec), and QTcF Interval (msec), by treatment and overall for subjects in the safety analysis set. Changes from baseline to each scheduled post-baseline visit will be presented.

All ECG data (both observed and change from baseline) will be presented in a listing.

#### 8.6. Other Safety Data

The site of study drug infusion will be evaluated for signs of infusion-related reactions on Day 1 at 15 minutes, 0.5-1.0 hours, and 3.0 hours ( $\pm$  15 minutes), and at the follow-up visit on Day 8 ( $\pm$ 1 day). Any reaction observed will be recorded in the CRF as an AE.

A summary table presenting observed values will be presented. All infusion site assessment data will be presented in a listing.

#### 9. Pharmacokinetics

Four PK blood collections will be obtained in a subset of approximately 40 subjects to determine the cefazolin plasma concentrations in this population. Pharmacokinetic samples will be obtained at 0.5 to 1.0 hours, 2.0 hours ( $\pm$  15 minutes), 3.0 hours ( $\pm$  15 minutes), and 4.0 hours ( $\pm$  15 minutes) after the start of the study drug infusion.

If the surgery is unexpectedly extended beyond the 3-hour limit and an additional dose of study drug will be administered best efforts will be made to obtain the 3-hour and possibly the 4-hour PK samples prior to administration of the additional dose of study drug. Pharmacokinetic sample collection will not continue after the administration of an additional dose of study drug. In the cases of an additional dose of study drug, subjects from whom a 3-hour PK sample is obtained prior to administration of the additional dose are considered PK completers.

Cefazolin plasma concentrations will be listed by subject and scheduled time point/interval. Concentrations will also be summarized by treatment and age bracket for each schedule time point/interval using descriptive statistics (n, mean, SD, % coefficient of variation, median, minimum, and maximum).

Mean cefazolin plasma concentrations versus scheduled time point/interval will be presented on linear and semi-logarithmic plots. Individual cefazolin plasma concentrations versus actual time point will be presented on linear and semi-logarithmic plots.

Cefazolin plasma concentrations will be used for population PK modeling. Details of the population PK model will be contained in a separate document.

#### 10. Interim Analysis

No interim analysis will be conducted in this study.

#### 11. References

Trang M, Forrest A, Rubino C. Population PK Analysis for Cefazolin Using Data from HC-G-H-1202: Implications for Dosing in Children, Report from Institute for Clinical Pharmacodynamics for B. Braun Medical Inc. 2014. 72 p.

# 12. Appendices

# 12.1. Schedule of Study Procedures

| Study Phase | Screening<br>Period | Treatment Period (Day of Surgery) | | | | | Follow-up<br>Period | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>1</sup> | Pre-<br>surgery | | | Surgery | | | Post-<br>surgery <sup>2</sup> | Safety<br>Follow-up<br>Visit <sup>3</sup> |
| Study Day | Up to 30 Days<br>Before Study<br>Drug<br>Administration | | | | 1 | | | 1 or 2 | 8 (±1) |
| Time point after start of infusion | | | 15<br>min<br>(±5<br>min<br>) | 0.5 h - 1.0<br>h | 2.0 h<br>(±15 min) | 3.0 h<br>(±15 min) | 4.0 h<br>(±15<br>min) | | |
| Informed consent for study participation | X | | | | | | | | |
| Informed consent for pharmacokinetic (PK) participation | X | | | | | | | | |
| Inclusion/exclusion criteria | X | | | | | | | | |
| Subject identification number assignment | X | | | | | | | | |
| Demographics | X | | | | | | | | |
| Height (without shoes) | X | | | | | | | | |
| Weight <sup>4</sup> | X | X | | | | | | | |
| Medical history | X | | | | | | | | |
| Medication history | X | | | | | | | | |

| Study Phase | Screening<br>Period | Treatment Period (Day of Surgery) | | | | | Follow-up<br>Period | | |
|---|---|---|---|---|---|---|---|---|---|
| Procedure | Screening <sup>1</sup> | surgery su | | | | Post-<br>surgery <sup>2</sup> | Safety<br>Follow-up<br>Visit <sup>3</sup> | | |
| Study Day | Up to 30 Days<br>Before Study<br>Drug<br>Administration | | | | | 1 or 2 | 8 (±1) | | |
| Time point after start of infusion | | | 15<br>min<br>(±5<br>min<br>) | 0.5 h - 1.0<br>h | 2.0 h<br>(±15 min) | 3.0 h<br>(±15 min) | 4.0 h<br>(±15<br>min) | | |
| Updated medical history for eligibility | | X | | | | | | | |
| Physical examination <sup>5</sup> | X | X | | | | | | X | X |
| Vital signs <sup>6, 7</sup> | X | $X^7$ | X | X | | X | | X | X |
| Electrocardiograph (ECG) <sup>6</sup> | X | | | | | | | X | |
| Clinical Laboratory tests (blood) <sup>8</sup> | X <sup>9</sup> | X | | | | | | X | X |
| Pregnancy test <sup>10</sup> | X | X | | | | | | | |
| Study drug infusion site assessment | | | X | X | | X | | X | X |
| Pharmacokinetic blood collection <sup>11</sup> | | | | X | X | X | X | | |
| Concomitant medications | | | • | • | Continuous | | | | • |
| Adverse event monitoring | | | | | Continuous | | | | |
| Study drug administration <sup>12</sup> | | X | | | | | | | |

- <sup>1</sup> If Screening visit occurs on Day 1 (day of surgery), all Screening visit assessments must be properly completed.
- Postsurgery assessments will be performed at 24 hours after surgery or discharge from the study site, whichever comes first.
- Safety Follow-up visit will be performed for subjects who complete the study or terminate prematurely after receiving study drug, whenever possible.
- Weight will be measured with indoor clothing and without shoes.
- Details of physical examination are outlined in Section 6.2.2 of the protocol. The complete physical examination includes an assessment of general appearance and a review of systems (dermatologic, head, eyes, ears, nose, mouth/throat/neck, thyroid, lymph nodes, and respiratory, cardiovascular, gastrointestinal, extremities, musculoskeletal, neurologic, and psychiatric systems). A brief physical examination will be performed both before and after dosing on Day 1 and at the Safety Follow-up visit.
- Vital signs (including blood pressure [systolic and diastolic], pulse, body temperature, and respiratory rate) and ECGs should be taken with subjects in supine position after resting for 5 minutes. Details of vital sign measurements are outlined in Section 6.2.3 of the protocol. Details of ECGs are outlined in Section 6.2.4 of the protocol. Vital signs and ECG obtained at Screening will be considered as Baseline.
- <sup>7</sup> Predose vital sign measurements should be obtained within approximately 30 minutes before the start of study drug administration.
- <sup>8</sup> Clinical laboratory tests will include hematology and clinical chemistry. Details of laboratory tests are outlined in Section 6.4 of the protocol. Laboratory tests except for screening procedures will be performed by the central laboratory.
- Screening laboratory tests should be performed within 30 days of Day 1 and can be the same tests as those assessed for surgical clearance. Screening laboratory tests will be performed at local laboratories.
- Urine pregnancy tests will be performed for all females of childbearing potential at Screening and be repeated on Day 1. If positive, pregnancy will be confirmed with serum test. If pregnancy is confirmed, the subject will not be enrolled or if already enrolled and not yet dosed the subject will be dropped. If a pregnant subject is administered study drug in error, the subject will be followed through the completion or termination of the pregnancy. All pregnancy tests will be performed at local laboratories.
- Pharmacokinetic blood samples will be obtained at the designated time points after the <u>start</u> of the study drug infusion. NOTE: The catheter that is used for study drug infusion and the arm it is inserted in cannot be used for collection of the PK samples. Pharmacokinetic samples must be taken from the opposite arm of the study drug infusion.
- Study drug will be administered over 30 minutes as an infusion starting 0.5 to 1 hour before surgery begins and following institutional guidelines. The start time of the study drug infusion and the start time of the anesthesia induction will be recorded in the CRF. Subjects with a weight of at least 25 kg but less than 60 kg will receive 1-g cefazolin. Subjects with a weight of at least 60 kg will receive 2-g cefazolin. If the surgery is extended unexpectedly beyond the 3-hour limit, additional doses of study drug are permitted according to institutional guidelines.

# 12.2. Table, Listing, and Figure Shell Table of Contents

# **Tables**

| Table 14.1.1 | Subject Disposition (Safety Analysis Set) |
|---|---|
| Table 14.1.2.1 | Demographic and Baseline Characteristics (Safety Analysis Set) |
| Table 14.1.2.1 | Demographic and Baseline Characteristics (Pharmacokinetic |
| | Analysis Set) |
| Table 14.2.1.1 | Summary of Plasma Concentrations of Cefazolin by Treatment and |
| | Age (Pharmacokinetic Analysis Set) |
| Table 14.3.1.1 | Overall Summary of Adverse Events (Safety Analysis Set) |
| Table 14.3.1.2 | Adverse Events (Safety Analysis Set) |
| Table 14.3.1.3 | Adverse Events by Relationship to Study Drug (Safety Analysis Set) |
| Table 14.3.1.4 | Adverse Events by Severity (Safety Analysis Set) |
| Table 14.3.4.1 | Summary and Change from Baseline in Hematology (Safety Analysis Set) |
| Table 14.3.4.2 | Summary and Change from Baseline in Clinical Chemistry (Safety |
| T 11 1405 | Analysis Set) |
| Table 14.3.5 | Summary and Change from Baseline in Vital Sign Measurements |
| T 11 1426 | (Safety Analysis Set) |
| Table 14.3.6 | Summary and Change from Baseline in Electrocardiograms (Safety Analysis Set) |
| Table 14.3.7 | Summary of Infusion Site Assessments (Safety Analysis Set) |
| Listings | |
| J | Subject Disposition |
| Listings Listing 16.2.1.1 Listing 16.2.1.2 | Subject Disposition Informed Consent and Assent |
| Listing 16.2.1.1<br>Listing 16.2.1.2 | • |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1 | Informed Consent and Assent |
| Listing 16.2.1.1<br>Listing 16.2.1.2 | Informed Consent and Assent<br>Admission Criteria Deviations<br>Protocol Deviations |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2 | Informed Consent and Assent<br>Admission Criteria Deviations<br>Protocol Deviations<br>Subjects Excluded from Analysis Sets |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3 | Informed Consent and Assent<br>Admission Criteria Deviations<br>Protocol Deviations |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3<br>Listing 16.2.4.1 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3<br>Listing 16.2.4.1<br>Listing 16.2.4.2<br>Listing 16.2.4.3 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3<br>Listing 16.2.4.1<br>Listing 16.2.4.2 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.3 Listing 16.2.4.4 Listing 16.2.4.5 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery |
| Listing 16.2.1.1<br>Listing 16.2.1.2<br>Listing 16.2.2.1<br>Listing 16.2.2.2<br>Listing 16.2.3<br>Listing 16.2.4.1<br>Listing 16.2.4.2<br>Listing 16.2.4.3<br>Listing 16.2.4.4 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.3 Listing 16.2.4.5 Listing 16.2.5 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery Study Drug Administration |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.4 Listing 16.2.4.5 Listing 16.2.5 Listing 16.2.6.1 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery Study Drug Administration Individual Plasma Concentrations of Cefazolin |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.4 Listing 16.2.4.5 Listing 16.2.5 Listing 16.2.5 Listing 16.2.7.1 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery Study Drug Administration Individual Plasma Concentrations of Cefazolin Adverse Events Serious Adverse Events |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.3 Listing 16.2.4.5 Listing 16.2.5 Listing 16.2.5 Listing 16.2.7.1 Listing 16.2.7.2 Listing 16.2.7.3 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery Study Drug Administration Individual Plasma Concentrations of Cefazolin Adverse Events Serious Adverse Events Adverse Events Leading to Early Discontinuation |
| Listing 16.2.1.1 Listing 16.2.1.2 Listing 16.2.2.1 Listing 16.2.2.2 Listing 16.2.3 Listing 16.2.4.1 Listing 16.2.4.2 Listing 16.2.4.3 Listing 16.2.4.3 Listing 16.2.4.5 Listing 16.2.5 Listing 16.2.5 Listing 16.2.7.1 Listing 16.2.7.2 | Informed Consent and Assent Admission Criteria Deviations Protocol Deviations Subjects Excluded from Analysis Sets Demographic and Baseline Characteristics Medical History Prior and Concomitant Medications Medical and Surgical Treatment Procedures Surgery Study Drug Administration Individual Plasma Concentrations of Cefazolin Adverse Events Serious Adverse Events |

| Listing 16.2.8.3 | Pregnancy Test Results |
|---|---|
| Listing 16.2.9.1 | Vital Sign Measurements |
| Listing 16.2.9.2 | Electrocardiograms |
| Listing 16.2.9.3 | Abnormal Physical Examination Findings |
| Listing 16.2.9.4 | Infusion Site Assessments |
| Figures | |
| <b>Figures</b> Figure 14.2.1 | Mean (+/-SD) Plasma Concentrations of Cefazolin versus Time |
| 3 | Mean (+/-SD) Plasma Concentrations of Cefazolin versus Time (Pharmacokinetic Analysis Set) |
| 3 | |

Table 14.1.1 Subject Disposition Safety Analysis Set

| | Treatment A | Treatment B | Total |
|------------------------------------|-------------|-------------|-----------|
| | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (%) | n (%) |
| Total Number of Subjects | | | |
| Completed | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Discontinued | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Primary Reason for Discontinuation | | | |
| Protocol violation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Noncompliance with the protocol | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Serious AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Intolerable AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Lost to follow-up | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Pregnancy | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Subject withdrew consent | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| LAR withdrew consent [1] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Investigator decision | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Analysis Sets | | | |
| Safety [2] | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PK [3] | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: Percentages are based on the number of subjects in the safety analysis set.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.1 and Listing 16.2.3

<sup>[1]</sup> LAR = Legally Authorized Representative.

<sup>[2]</sup> Safety analysis set includes all subjects who received any study drug.
[3] Pharmacokinetic (PK) analysis set includes all subjects from whom at least one measurable concentration PK sample

Table 14.1.2.1
Demographic and Baseline Characteristics
Safety Analysis Set

| | Treatment A | Treatment B | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=XX) |
| Age (years) | | | |
| n | XX | XX | XX |
| Mean (SD) | xx.x (x.xx) | xx.x (x.xx) | xx.x (x.xx) |
| Median | XX.X | xx.x | XX.X |
| Min, Max | XX, XX | XX, XX | xx, xx |
| Age categories, n (%) | | | |
| >=10 to <=13 years | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| >13 to <=17 years | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Sex, n (%) | | | |
| Female | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Male | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Race, n (%) | | | |
| White | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Black or African American | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Asian | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| American Indian or Alaska Native | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Native Hawaiian or Other Pacific Islander | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Multi-racial | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Ethnicity, n (%) | | | |
| Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Not Hispanic or Latino | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to programmer: Summarize subjects who report two or more races as "Multi-racial". If there are no such subject, remove "Multi-racial" category. Continue with Height (cm) and Weight (kg)

Note: Percentages are based on the number of subjects in the safety analysis set.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.4.1

Table 14.1.2.2

Demographic and Baseline Characteristics
Pharmacokinetic Analysis Set

Use the same Table shell as for Table 14.1.2.1, but display for the PK analysis set. Source Data: Listing 16.2.4.1

Table 14.2.1.1

Summary of Plasma Concentrations of Cefazolin by Treatment and Age
Pharmacokinetic Analysis Set

| | | Treatment A | | | Treatment B | | |
|---|---|---|---|---|---|---|---|
| Scheduled | | >=10 to <=13 | >13 to <=17 | | >=10 to <=13 | >13 to <=17 | |
| Time Point | Statistics | years old | years old | All Ages | years old | years old | All Ages |
| 0.5-1.0 HR | n | XX | XX | XX | XX | XX | XX |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XXX | xx.xxx | XX.XXX | XX.XXX | XX.XXX | XX.XXX |
| | CV% | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Median | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Min | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |
| | Max | XX.X | XX.X | XX.X | XX.X | XX.X | XX.X |

Note to Programmer: Sort by Scheduled Time Point. Plasma samples for PK assessments of Cefazolin will be collected from all subjects at the following time points: between 0.5-1 hr, 2, 3, and 4 hr relative to start of study drug infusion. Concentrations that are BLQ will be treated as 0. Mean BLQ concentrations will be presented as 0, SD and CV will be presented as NA.

Note: Concentrations that were BLQ were treated as zero for descriptive statistics. NA = Not applicable. Sample collection times are from the start of infusion.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.6.1.

Table 14.3.1.1 Overall Summary of Adverse Events Safety Analysis Set

| | Treatment A (N=xx) n (%) | Treatment B (N=xx) n (%) | Total (N=xx) n (%) |
|---|---|---|---|
| Any AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Treatment-Related AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Moderate AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Treatment-Related Moderate AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Severe AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Treatment-Related Severe AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any SAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Treatment-Related SAE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any AE Leading to Early Discontinuation | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Any Death | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note: A treatment-related AE is defined as any AE with a relationship designated as 'Possible', 'Probable', or 'Definite' by the investigator. At each level of subject summarization, a subject is counted once if the subject reported one or more events. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the safety analysis set within each treatment and overall.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.7.1, Listing 16.2.7.2 and Listing 16.2.7.3

Table 14.3.1.2 Adverse Events Safety Analysis Set

| | Treatment A | Treatment B | Total |
|----------------------|-------------|-------------|-----------|
| System Organ Class | (N=xx) | (N=xx) | (N=xx) |
| Preferred Term | n (%) | n (%) | n (%) |
| All AE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to Programmer: System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no AEs, then display "No adverse events were reported."

Note: At each level of subject summarization, a subject is counted once if the subject reported one or more events. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the safety analysis set within each treatment and overall. Adverse events were coded using MedDRA version 19.1.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.7.1

Table 14.3.1.3

Adverse Events by Relationship to Study Drug

Safety Analysis Set

| System Organ Class | Treatment A | Treatment B | Total |
|----------------------|-------------|-------------|-----------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| Relationship | n (%) | n (%) | n (%) |
| All AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| UNRELATED | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| POSSIBLE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PROBABLE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| DEFINITE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| UNRELATED | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| POSSIBLE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| PROBABLE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| DEFINITE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to programmer: System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no AEs, then display "No adverse events were reported."

Note: At each level of subject summarization, a subject is counted once for the most related event. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety analysis set within each treatment and overall. Adverse events were coded using MedDRA version 19.1.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.7.1

Table 14.3.1.4

Adverse Events by Severity
Safety Analysis Set

| System Organ Class | Treatment A | Treatment B | Total |
|----------------------|-------------|-------------|-----------|
| Preferred Term | (N=xx) | (N=xx) | (N=xx) |
| Relationship | n (%) | n (%) | n (%) |
| All AEs | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MILD | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MODERATE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SEVERE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| System Organ Class 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MILD | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| MODERATE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| SEVERE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 1 | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Preferred Term 2 | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to programmer: System organ class is displayed in descending order of frequency for "Total" then alphabetically. Preferred term is displayed in descending order of frequency for "Total" then alphabetically within system organ class. If there are no AEs, then display "No adverse events were reported."

Note: At each level of subject summarization, a subject is counted once for the most severe event. n represents the number of subjects at each level of summarization. Percentages are based on the number of subjects in the Safety analysis set within each treatment and overall. Adverse events were coded using MedDRA version 19.1.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.7.1

B. Braun Medical Inc. Protocol: HC-G-H-1601

Table 14.3.4.1

Summary and Change from Baseline in Hematology
Safety Analysis Set

Parameter (Unit): XXXXXXXXXX (XXXX)

| Visit | Actua | | | Actual Value | | Change from Baseline | | | ne | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Treatment B (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Postsurgery | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Treatment B (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |

Note to programmer: The post-baseline visits are: Postsurgery, and Follow-up. Start a new page for each parameter.

Note: Baseline is defined as the screening visit; Postsurgery is defined as 24 hours after surgery or at discharge from the study site, whichever comes first.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.8.1

Table 14.3.4.2
Summary and Change from Baseline in Clinical Chemistry
Safety Analysis Set

Use the same Table shell as for Table 14.3.4.1, but display Clinical Chemistry parameters. Source Data: Listing 16.2.8.2

Parameter (Unit): XXXXXXXXXX (XXXX)

| Visit/Timepoint | | | Actual V | Value | | | Change from Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Treatment B (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Day 1/Pre-dose | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Treatment B (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |

Note to programmer: The post-baseline visit/timepoints are: Day 1/Pre-dose, Day 1/15 min, Day 1/.5hr-1.0hr, 3.0hr, Postsurgery, and Follow-up. Start a new page for each parameter.

Note: Baseline is defined as the screening visit.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.9.1

 $\begin{array}{c} \text{Table 14.3.6} \\ \text{Summary and Change from Baseline in Electrocardiograms} \\ \text{Safety Analysis Set} \end{array}$ 

Parameter (Unit): XXXXXXXXXX (XXXX)

| Visit | | | Actual ' | Value | | | Change from Baseline | | | ie | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Treatment | n | Mean | SD | Median | Min | Max | n | Mean | SD | Median | Min | Max |
| Baseline | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Treatment B (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | | | | | | |
| Postsurgery | | | | | | | | | | | | |
| Treatment A (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Treatment B (N=xx) | XX | XX.X | XX.XX | xx.x | XX | XX | XX | XX.X | XX.XX | XX.X | XX | XX |
| Total (N=xx) | XX | XX.X | XX.XX | XX.X | XX | XX | XX | XX.X | xx.xx | XX.X | XX | XX |

Note to programmer: The post-baseline visits are: Postsurgery and Follow-up. Start a new page for each parameter.

Note: Baseline is defined as the screening visit.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.9.2

Table 14.3.7
Summary of Infusion Site Assessments
Safety Analysis Set

| Visit/Timepoint | Treatment A | Treatment B | Total |
|---------------------|-------------|-------------|-----------|
| Assessment | (N=xx) | (N=xx) | (N=xx) |
| Response | n (%) | n (%) | n (%) |
| Day 1/15 min | | | |
| Pain | | | |
| YES | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOT DONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Erythema/Redness | | | |
| YES | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOT DONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Induration/Swelling | | | |
| YES | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOT DONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Localized Warmth | | | |
| YES | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOT DONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| Other | | | |
| YES | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NO | xx (xx.x) | xx (xx.x) | xx (xx.x) |
| NOT DONE | xx (xx.x) | xx (xx.x) | xx (xx.x) |

Note to programmer: The visit/timepoints are: Day 1/15 min, Day 1/.5hr-1.0hr, 3.0hr, Postsurgery, and Follow-up. Present the Assessments in the order shown (Pain, Erythema/Redness, Induration/Swelling, Localized Warmth, and Other).

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.9.4

# Listing 16.2.1.1 Subject Disposition

Treatment: A

| Date of | | Date (Day) of | Completed | Discontinuation | |
|---|---|---|---|---|---|
| Subject | Dose | Final Contact | Study? | Date (Day) | Reason |
| xxxxxx | DDMMMYYYY | DDMMMYYYY (xx) | Yes | | |
| xxxxxxx | DDMMMYYYY | DDMMMYYYY (xx) | No | DDMMMYYYY (xx) | xxxxxxxxxx |
| xxxxxx | DDMMMYYYY | DDMMMYYYY (xx) | No | DDMMMYYYY (xx) | Adverse Event: xxxxx |

Note to Programmer: Sort by treatment and subject. If discontinuation occurred due to AE, append the corresponding AE term. Start a new page for each treatment.

Note: Day corresponds to study day. Day 1 is date of surgery.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Listing 16.2.1.2
Informed Consent and Assent

Treatment: A

| | | | | Pharmacokinetic (PK) Blood Collection | | |
|---|---|---|---|---|---|---|
| Subject | Informed<br>Consent Date | HIPAA<br>Auth.<br>Date | Assent Required?/ Assent Date | Did subject consent to participate in PK sampling? | PK Informed<br>Consent Date | PK Assent<br>Required?/<br>PK Assent Date |
| xxxxxxx | DDMMMYYYY | DDMMMYYYY | Yes/<br>DDMMMYYYY | Yes | DDMMMYYYY | No |
| xxxxxx | DDMMMYYYY | DDMMMYYYY | Yes/<br>DDMMMYYYY | Yes | DDMMMYYYY | Yes/<br>DDMMMYYYY |
| xxxxxx | DDMMMYYYY | DDMMMYYYY | No | No | | |

Note to Programmer: Sort by treatment and subject. If discontinuation occurred due to AE, append the corresponding AE term. Start a new page for each treatment.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.
Listing 16.2.2.1
Admission Criteria Deviations

Treatment: x

| Subject | Protocol Date - Version | Criteria Type | Criteria Number | Comment |
|---|---|---|---|---|
| xxxxxx | DDMMMYYYY - xxxxxxx | Inclusion | xx | |
| xxxxxxx | DDMMMYYYY - xxxxxx | Exclusion | xx | |

•••

Note to Programmer: Sort by treatment and subject. Start a new page for each treatment. If there are no admission criteria deviations, then display "No admission criteria deviations were reported."

#### Deviated criteria:

Inclusion xx: xxxxxxxxxxxxxxxxxxxxx

Exclusion xx: xxxxxxxxxxxxx

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

# Listing 16.2.2.2 Protocol Deviations

Treatment: x

| Subject | Date (Day) [1]<br>of Deviation | Deviation Type | Description |
|---------|--------------------------------|----------------|--------------|
| xxxxxx | DDMMMYYYY (xx) | xxxxxxxx | xxxxxxxxxxxx |
| xxxxxx | DDMMMYYYY (xx) | xxxxxxxx | xxxxxxxxxxxx |

Note to Programmer: Sort by treatment and subject. Start a new page for each treatment. If there are no protocol deviations, then display "No protocol deviations were reported."

<sup>[1]</sup> Day corresponds to study day. Day 1 is date of surgery.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

B. Braun Medical Inc. Protocol: HC-G-H-1601

# Listing 16.2.3 Subjects Excluded from Analysis Sets

Treatment: x

| Subject | Excluded from Safety [1]/<br>Reason for Exclusion | Excluded from Pharmacokinetic [2]/<br>Reason for Exclusion |
|---|---|---|
| xxxxxx | No | Yes/<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |
| xxxxxx | No | No |
| XXXXXXX | Yes/<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx | Yes/<br>xxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxxx |

Note to Programmer: Sort by treatment and subject. Start a new page for each treatment.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

<sup>[1]</sup> Safety analysis set includes all subjects who received any study drug.

<sup>[2]</sup> Pharmacokinetic (PK) analysis set includes all subjects from whom at least one measurable concentration PK sample is obtained.

Listing 16.2.4.1
Demographic and Baseline Characteristics

Treatment: A

| | | Age | | | | Scre | ening |
|---|---|---|---|---|---|---|---|
| | | (years) | | | Eth. | Height | Weight |
| Subject | Date of Birth | [1] | Sex | Race | [2] | (cm) | (kg) |
| xxxxxx | DDMMMYYYY | XX | Male | xxxxxxxxxxxx | Н | XXX.X | XXX.X |
| xxxxxx | DDMMMYYYY | XX | Female | xxxxxxxx | N | xxx.x | xx.x |
| xxxxxx | DDMMMYYYY | XX | xxxxxx | xxxxxxxxxx | X | xxx.x | xxx.x |

Note to Programmer: Sort by treatment and subject. Start a new page for each treatment.

<sup>[1]</sup> Age in years is the integer part of (Date of Informed Consent - Date of Birth)/365.25.

<sup>[2]</sup> Ethnicity: H = Hispanic or Latino, N = Not Hispanic or Latino.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Listing 16.2.4.2 Medical History

Treatment: x

| Subject | Body System | Condition/Diagnosis | System Organ Class [1]/<br>Preferred Term [1] | Start/Stop<br>Date |
|---|---|---|---|---|
| xxxxxx | xxxxxxxxxxxxx | xxxxxxxx | xxxxxxxxxxxxxx/<br>xxxxxxxxxxx | DDMMMYYYY/<br>DDMMMYYYY |
| xxxxxx | xxxxxxxxxx | xxxxxxxxx | xxxxxxxxxxxxx/<br>xxxxxxxxxxxxxx | DDMMMYYYY/<br>Ongoing |

...

Note to Programmer: Sort by treatment, subject, condition/diagnosis, and start/stop date. Start a new page for each treatment. Display "Ongoing" in place of Stop Date if the condition is ongoing. If there are no medical histories, then display "No medical histories were reported."

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

<sup>[1]</sup> From MedDRA version 19.1.

Listing 16.2.4.3 Prior and Concomitant Medications

Treatment: x

| | | | | | | Start/Stop | | |
|---|---|---|---|---|---|---|---|---|
| | Med | Preferred Drug Name [1]/ | Type | | | Date (Day) [3]/ | Route/ | Indication |
| Subject | ID | Drug Name | [2] | Dose | Unit | Time | Frequency | (AE ID) |
| XXXXXXX | XXX | xxxxxxxxxxxx/ | PC | XXXX | XXXXXXX | DDMMMYYYY (xx)/ | xxxxxxx/ | XXXXXXXX |
| | | xxxxxxxxxxx | | | | HH:MM/ | xxxxxxxxx | |
| | | | | | | Ongoing | | |
| | XXX | xxxxxxxxxxxx/ | P | XX.X | XXXXXX | DDMMMYYYY (xx)/ | xxxxxxx/ | XXXXXXXXXX |
| | | xxxxxxxxxxx | | | | HH:MM/ | XXXXXXXXX | |
| | | | | | | DDMMMYYYY (xx)/ | | |
| | | | | | | HH:MM | | |
| | XXX | xxxxxxxxxxxx/ | С | XXXX | xxxxx | DDMMMYYYY (xx)/ | xxxxxxx/ | xxxxxxxx |
| | | xxxxxxxxxx | | | | HH:MM/ | XXXXXXXXX | (xxxx) |
| | | | | | | DDMMMYYYY (xx)/ | *************************************** | () |
| | | | | | | , , , | | |
| | | | | | | HH:MM | | |

Note to Programmer: Sort by treatment, subject, preferred drug name, and date/time started. Start a new page for each treatment. Display "Ongoing" in place of Stop Date/Time if the medication is ongoing. If there are no prior or concomitant medications, then display "No prior or concomitant medications were reported."

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

<sup>[1]</sup> From WHODrug version 01DEC2016.

<sup>[2]</sup> P = Prior, C = Concomitant.

<sup>[3]</sup> Day corresponds to study day. Day 1 is date of surgery.

Listing 16.2.4.4
Medical or Surgical Treatment Procedures

Treatment: x

| Subject | System Organ Class [1]/<br>Preferred Term [1]/<br>Procedure | Reason [AE ID] | Start/Stop<br>Date (Day) [2] |
|---|---|---|---|
| xxxxxx | ************************************** | xxxxxxxxxx [xxxxxxxx] | DDMMMYYYY (xx)/<br>DDMMMYYYY (xx) |
| xxxxxx | xxxxxxxxxxx/<br>xxxxxxxxxxxx/<br>xxxxxxxxxxx | Other: XXXXXXXX | DDMMMYYYY (xx)/<br>Ongoing |

•••

Note to Programmer: Sort by treatment, subject, procedure, and start/stop date. If procedure is ongoing then display "Ongoing" in the place of Stop Date. If the procedure was for an AE, please attach the corresponding AE ID to Reason. Start a new page for each treatment.

If there are no medical or surgical treatment procedures, then display "No medical or surgical treatment procedures were reported."

Treatment A: 1g cefazolin for pediatric surgical subjects weighing  $\geq$ = 25 kg but < 60 kg;

<sup>[1]</sup> From MedDRA, version 19.1.

<sup>[2]</sup> Day corresponds to study day. Day 1 is date of surgery.

Listing 16.2.4.5

Treatment: x

| Subject | Procedure | Start/Stop<br>Date/Time | Anesthesia Start<br>Date/Time | Comment |
|---|---|---|---|---|
| xxxxxx | xxxxxxxxxxxxxxxx | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM | xxxxxxxxxx |
| xxxxxx | xxxxxxxxxxx | DDMMMYYYYHH:MM/<br>MM:HH\YYYYMMDD | DDMMMYYYY/HH:MM | |

Surgery

...

Note to Programmer: Sort by treatment, subject, procedure, and start/stop date. Start a new page for each treatment.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Listing 16.2.5
Study Drug Administration

Treatment: x

| | | Lot Number/ | Dose | | Interrupt/ | |
|---|---|---|---|---|---|---|
| | Catheter | Reconstitution | Start/Stop | Volume | Restart | |
| Subject | Location [1] | Date/Time | Date/Time | (mL) | Date/Time | Comment |
| xxxxxx | RIGHT HAND | xxxxxxx/<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | xx | DDMMMYYYY/HH:MM/<br>DISCONTINUED | xxxxxxxxx |
| xxxxxx | LEFT FOREARM | xxxxxxx/<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | xx | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | xxxxxx |
| xxxxxx | RIGHT HAND | xxxxxxx/<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | xx | NOT INTERRUPTED | |
| | LEFT LEG S | xxxxxxx/<br>DDMMMYYYY/HH:MM | DDMMMYYYY/HH:MM/<br>DDMMMYYYY/HH:MM | xx | NOT INTERRUPTED | xxxxxxxx |

...

Note to programmer: Sort by treatment, subject, and start date/time. If study drug was not interrupted, display "NOT INTERRUPTED" in Interrupt/Restart Date/Time column. If drug was discontinued without restart, display 'DISCONTINUED' for Restart Date/Time. If record represents a supplemental infusion, display 'S' after Catheter Location.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

<sup>[1]</sup> S = Supplemental infusion.

Listing 16.2.6.1
Individual Plasma Concentrations of Cefazolin
Pharmacokinetic Analysis Set

Treatment: A

| Subject/ | | | Deviation from | | |
|---|---|---|---|---|---|
| Age (yr)/ | Scheduled | Sample Collection | Scheduled Time | Cefazolin | |
| Weight (kg) | Time | Date/Time | (minutes) | Concentration (unit) | Comment |
| xxxxxxx/xx/xx | 0.5-1.0 HR | DDMONYYYY/HH:MM | | XX.XX | xxxxxxxxxxx |
| | 2 HR | DDMONYYYY/HH:MM | X | XX.XX | |
| | 3 HR | DDMONYYYY/HH:MM | x | XX.XX | |
| | 4 HR | DDMONYYYY/HH:MM | X | XX.XX | |
| xxxxxxx/xx/xx | 0.5-1.0 HR | DDMONYYYY/HH:MM | | XX.XX | xxxxxxxxxxx |
| | 2 HR | DDMONYYYY/HH:MM | x | XX.XX | |
| | 3 HR | DDMONYYYY/HH:MM | x | XX.XX | |
| | 4 HR | DDMONYYYY/HH:MM | X | XX.XX | |
| xxxxxxx/xx/xx | 0.5-1.0 HR | DDMONYYYY/HH:MM | | XX.XX | xxxxxxxxxxx |
| | 2 HR | DDMONYYYY/HH:MM | X | XX.XX | |
| | 3 HR | DDMONYYYY/HH:MM | x | XX.XX | |
| | 4 HR | DDMONYYYY/HH:MM | X | XX.XX | |

Note: The lower limit of quantification is x.xx ng/mL for cefazolin. NS = no sample.

Sample collection times are from the start of infusion.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: CRF data and concentration data.

Note to Programmer: Sort by Subject and Schedule Time. Repeat for Treatment B. Plasma samples for PK assessments of Cefazolin will be collected from all subjects at the following time points: between 0.5-1 hr, 2, 3, and 4 hr relative to start of study drug infusion.

Listing 16.2.7.1
Adverse Events

Treatment: A

| Subject | AE<br>ID | System Organ Class/<br>Preferred Term/<br>Adverse Event | Start/Stop<br>Date (Day) [1]/<br>Time | Frequency/<br>Severity/<br>Relationship | Action/<br>Outcome/<br>Serious | Treatment<br>Required |
|---|---|---|---|---|---|---|
| xxxxxx | XX | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (xx)/<br>HH:MM<br>DDMMMYYYY (xx)/<br>HH:MM | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXX/<br>XXXXXXXX/<br>XX | XXXXXXX |
| xxxxxx | XX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (xx)/<br>HH:MM<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXXX/<br>XXXXXXXX/<br>XX | XXXXXXX |

...

Note to Programmer: Sort by treatment, subject, and AE ID. Start a new page for each treatment. Display "Ongoing" in place of Stop Date/Time if the AE is ongoing.

If there are no AEs, then display 'No adverse events were reported.'

Note: Adverse events were coded by system organ class and preferred term using MedDRA Version 19.1.

[1] Day corresponds to study day. Day 1 is date of surgery.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

### Listing 16.2.7.2 Serious Adverse Events

Treatment: A

| Subject | AE<br>ID | System Organ Class/<br>Preferred Term/<br>Adverse Event | Start/Stop<br>Date (Day) [1]/<br>Time | Frequency/<br>Severity/<br>Relationship | Action/<br>Outcome/<br>Category [2] | Treatment<br>Required |
|---|---|---|---|---|---|---|
| xxxxxx | XX | XXXXXXXXXXXXXX/<br>XXXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (xx)/<br>HH:MM<br>DDMMMYYYY (xx)/<br>HH:MM | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXX/<br>XXXXXXXX/<br>XX | XXXXXX |
| xxxxxx | XX | XXXXXXXXXXXXXXX/<br>XXXXXXXXXXXXX/<br>XXXXXXXX | DDMMMYYYY (xx)/<br>HH:MM<br>Ongoing | XXXXXXXXX/<br>XXXXXXXXX/<br>XXXXXXXXX | XXXXXXXX/<br>XXXXXXX/<br>XX | xxxxxx |

Note to Programmer: Sort by treatment, subject, and AE ID. Start a new page for each treatment. Display "Ongoing" in place of Stop Date/Time if the AE is ongoing.

If there are no AEs, then display 'No adverse events were reported.'

Note: Adverse events were coded by system organ class and preferred term using MedDRA Version 19.1.

- [1] Day corresponds to study day. Day 1 is date of surgery.
- [2] 1=Death, 2=Life Threatening, 3=Persistent or significant incapacity, 4=Congenital anomaly or birth defect, 5=Hospitalization, 6=Prolonged Hospitalization, 7=Other important medical events

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Listing 16.2.7.3

Adverse Events Leading to Early Discontinuation

Use the same Listing shell as Listing 16.2.7.1, but display only AEs given on the study completion page when the primary reason for discontinuation was either Serious AE or Intolerable AE.

Listing 16.2.8.1 Hematology Laboratory Test Results

Treatment: x

| | | | Collection | | | | |
|---|---|---|---|---|---|---|---|
| | Lab Test | Visit | Date (Day) [2]/ | | Reference | Abnormal | |
| Subject | (Unit) | [1] | Time | Result | Range | Flag | Comment |
| xxxxxx | xxxxxxxxxxx<br>(xxxxx) | SCREENING | DDMONYYYY (xx)/<br>HH:MM | xxx.x | xxx.x - xxx.x | LOW | xxxxxxxxx |
| | | SCREENING, R | DDMONYYYY (xx)/<br>HH:MM | xxx.x | xxx.x - xxx.x | | xxxxxxx |
| | | ENROLLMENT | DDMONYYYY (xx)/<br>HH:MM | xxx.x | xxx.x - xxx.x | XXXX | |
| | | POSTSURGERY | DDMONYYYY (xx)/<br>HH:MM | XXX.X | xxx.x - xxx.x | | |

Note to Programmer: Sort by treatment, subject, lab test, and collection date/time. Start a new page for each treatment.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

<sup>[1]</sup> R = Repeat.

<sup>[2]</sup> Day corresponds to study day. Day 1 is date of surgery.

Listing 16.2.8.2 Clinical Chemistry Laboratory Test Results

Use the same Listing shell as Listing 16.2.8.1, but display clinical chemistry results.

Listing 16.2.8.3
Pregnancy Test Results

Treatment: x

| | Was Urine<br>Pregnancy | | Collection<br>Date (Day) [1]/ | | Serum Test |
|---|---|---|---|---|---|
| Subject | Performed? | Visit | Time | Result | Result [2] |
| xxxxxx | Yes | SCREENING | DDMONYYYY (xx)/ | Negative | |
| | | | HH:MM | | |
| | | ENROLLMENT | DDMONYYYY (xx)/ | Positive | Positive |
| | | | HH:MM | | |

...

Note to Programmer: Sort by treatment, subject, and collection date/time. Start a new page for each treatment. Only include females of childbearing potential.

[1] Day corresponds to study day. Day 1 is date of surgery.

[2] If urine test is positive, then a serum test is done for confirmation.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

## Listing 16.2.9.1 Vital Sign Measurements

Treatment: x

| Collection | | | Actual Value | | | | Change from Baseline [2] | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Visit/<br>Timepoint | Date (Day) [ | [1]/ | Body<br>Position | Sys<br>BP | Dia<br>BP | Pulse | Resp | Temp | Sys<br>BP | Dia<br>BP | Pulse | Resp | Temp |
| xxxxxx | SCREENING | DDMONYYYY (x: | (x)/ | SITTING | xxx | XX | XX | XX | xx.x | | | | | |
| | DAY 1/<br>PREDOSE | DDMONYYYY (x:<br>HH:MM | (x)/ | xxxxx | XXX | XX | XX | XX | xx.x | XXX | XX | XX | XX | XX.X |
| | DAY 1/<br>15 min | DDMONYYYY (x: HH:MM | (x)/ | xxxxxx | XXX | XX | XX | XX | XX.X | XXX | XX | XX | XX | XX.X |

Note to programmer: The post-baseline visits are: Day 1/Pre-dose, Day 1/15 min, Day 1/.5hr-1.0hr, 3.0hr, Postsurgery, and Follow-up. Start a new page for each treatment.

Note: Sys BP = Systolic Blood Pressure in mmHq; Dia BP = Diastolic Blood Pressure in mmHq; Pulse = Pulse in beats/min; Resp = Respiratory Rate in breaths/min; Temp = Temperature in degrees C.

[1] Day corresponds to study day. Day 1 is date of surgery.

[2] Baseline is defined as the screening visit.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Listing 16.2.9.2 Electrocardiograms

Treatment: x

| Collection<br>Date (Day)[1]/ | | Actual Value | | | | Change from Baseline [2] | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject | Visit | Time | HR | PR | QRS | QΤ | QTCF | Interpretation | HR | PR | QRS | QΤ | QTcF |
| xxxxxx | SCREENING | DDMONYYYY (xx)/<br>HH:MM | XXX | XX | XX | XXX | XXX | Normal | | | | | |
| | POSTSURGERY | DDMONYYYY (xx)/<br>HH:MM | XXX | XX | XX | XXX | XXX | xxxxxxxx | XXX | XX | XX | XX | XX |
| | FOLLOW=UP | DDMONYYYY (xx)/<br>HH:MM | XXX | XX | XX | XXX | XXX | xxxxxxx | XXX | XX | XX | XX | XX |

Note to programmer: The post-baseline visits are: Postsurgery and Follow-up. Start a new page for each treatment.

Note: HR = Heart rate in beats/min; PR = PR interval in msec; QRS = QRS duration in msec; QT = QT interval in msec; QTcF = QTcF interval in msec.

[1] Day corresponds to study day. Day 1 is date of surgery.

[2] Baseline is defined as the screening visit.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

B. Braun Medical Inc. Protocol: HC-G-H-1601

Listing 16.2.9.3
Abnormal Physical Examination Findings

Treatment: x

| Subject | Visit | Date (Day) [1] | Assessment | Findings |
|---|---|---|---|---|
| xxxxxx | SCREENING | DDMONYYYY (xx) | GENERAL APPEARANCE<br>DERMATOLOGIC<br>HEEN | xxxxxxxxxxxx |
| | POSTSURGERY | DDMONYYYY (xx) | <br>OVERALL | |

Note to Programmer: Sort by treatment, subject, date, and assessment (in the order as they appear in CRF with 'OVERALL' sorted last). Start a new page for each treatment. Include only those physical examinations with determined to be abnormal

[1] Day corresponds to study day. Day 1 is date of surgery.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Listing 16.2.9.4 Infusion Site Assessments

Treatment: x

| | | Date (Day) | | _ | |
|---|---|---|---|---|---|
| Subject | Visit/Timepoint | [1]/Time | Assessment | Result | Comment |
| xxxxxx | SCREENING | DDMONYYYY (xx)/<br>HH:MM | PAIN | YES | Xxxxxxx |
| | | | ERYTHEMA/REDNESS | NOT DONE | XXXXXXXXXXXXX |
| | | | INDURATION/SWELLING | NO | |
| | | | LOCALIZED WARMTH | NO | |
| | | | OTHER: XXXXXXX | NO | |
| | DAY 1/15 MIN | DDMONYYYY (xx)/<br>HH:MM | PAIN | YES | Xxxxxxx |
| | ••• | | | | |

Note to Programmer: Sort by treatment, subject, date/time, and assessment (in the order PAIN, ERYTHEMA/REDNESS, INDURATION/SWELLING, LOCALIZED WARMTH, OTHER). If OTHER, SPECIFY value is present, display "OTHER: xxxx" where "xxxx" is the value specified; otherwise display "OTHER". Start a new page for each treatment.

<sup>[1]</sup> Day corresponds to study day. Day 1 is date of surgery.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg;

Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Figure 14.2.1
Mean (+/-SD) Plasma Concentrations of Cefazolin versus Time
Pharmacokinetic Analysis Set

Age Bracket: >=10 to <=13 years old

Linear Scale



Semi-Logarithmic Scale



Note to programmer: Show both treatments on the same plot. Show treatments in legend. Repeat for age bracket >13 to  $\leq$ 17 years old and All Ages. Use the mid-point for the interval 0.5-1.0 hr for the x-axis coordinate.

Note: Concentrations that were BLQ were treated as zero for descriptive statistics. Sample collection times are from the start of infusion.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing  $\geq$  25 kg but < 60 kg; Treatment B: 2g cefazolin for pediatric surgical subjects weighing  $\geq$  60 kg.

Source Data: Table 14.2.1.1

Figure 14.2.2
Individual Plasma Concentrations of Cefazolin versus Time
Pharmacokinetic Analysis Set
Subject: xxxx
Age Bracket: xxxx

Linear Scale



Semi-Logarithmic Scale



Note to programmer: Show treatments in legend, same designations as F14.2.1.1. Set the y-axis scale uniform for each dose level.

Sample collection times are from the start of infusion.

Treatment A: 1g cefazolin for pediatric surgical subjects weighing >= 25 kg but < 60 kg; Treatment B: 2g cefazolin for pediatric surgical subjects weighing >= 60 kg.

Source Data: Listing 16.2.6.1